CLINICAL TRIAL: NCT00406640
Title: A Multicenter, Randomized, 8-Week Double-Blind Acute Phase Followed By a 6-Month Continuation Phase (Open-Label Or Double-Blind) Study to Evaluate the Efficacy, Safety, and Tolerability of DVS SR Versus Escitalopram in Postmenopausal Women With Major Depressive Disorder
Brief Title: Study Evaluating Desvenlafaxine Succinate Sustained Release (DVS SR) vs. Escitalopram in Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 3151A1-402
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Results first posted 2010-06-29 (Estimated); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Depression; Depressive Disorder; Depressive Disorder, Major
Keywords: MDD; Major Depressive Disorder; Depression
MeSH Terms: conditions — Depression; Depressive Disorder; Depressive Disorder, Major | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Desvenlafaxine succinate sustained-release (DVS SR)
- B (Active Comparator)
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Desvenlafaxine succinate sustained-release (DVS SR) — flexible dose of DVS 50-100 or 200 mg every day during 56 days. Extension until 6 months.
  Arms: A
Drug: Escitalopram — Flexible dose of Escitalopram 10 or 20 mg every day during 56 days. Extension until 6 months.
  Arms: B

SUMMARY:
Desvenlafaxine succinate (DVS) is a potent and selective serotonin and norepinephrine reuptake inhibitor (SNRI). This study will investigate the safety, efficacy, and tolerability of DVS SR versus escitalopram in women with major depressive disorder (MDD) who are postmenopausal.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women between the ages of 40 and 70 years, inclusive.
* A primary diagnosis of MDD, single or recurrent episode, without psychotic features using the modified MINI International Neuropsychiatric Interview (MINI).
* Montgomery-Asberg Depression Rating Scale (MADRS) total score > or = 22 at the screening and baseline visit.

Exclusion Criteria:

* Use of oral estrogen-, progestin-, androgen-, or Selective Estrogen Receptor Modulator (SERM)-containing drug products 8 weeks before baseline.
* Current (within 12 months) psychoactive substance abuse or dependence (including alcohol), manic episode, post-traumatic stress disorder, obsessive-compulsive disorder, or a lifetime diagnosis of bipolar or psychotic disorder.
* A history or active presence of clinically important medical disease.

Additional criteria apply.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 595 (Actual)
Dates: Start 2006-12; Primary Completion 2008-02 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Argentina: Scheima@wyeth.com; Trial Manager, Principal Investigator — For Chile: scheima@wyeth.com; Trial Manager, Principal Investigator — For Mexico: gomezzlj@wyeth.com
Locations (61):
- United States (49):
  - Peoria, Arizona
  - Pasadena, California
  - San Diego, California
  - Denver, Colorado
  - Cromwell, Connecticut
  - Farmington, Connecticut
  - Waterbury, Connecticut
  - Brooksville, Florida
  - Coral Springs, Florida
  - Fort Myers, Florida
  - Gainesville, Florida
  - Maitland, Florida
  - Atlanta, Georgia
  - Roswell, Georgia
  - Northfield, Illinois
  - Oak Brook, Illinois
  - Overland Park, Kansas
  - Wichita, Kansas
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Fall River, Massachusetts
  - Saint Paul, Minnesota
  - Las Vegas, Nevada
  - Piscataway, New Jersey
  - Elmsford, New York
  - Hollis, New York
  - New York, New York
  - Syracuse, New York
  - Raleigh, North Carolina
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - East Providence, Rhode Island
  - Lincoln, Rhode Island
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Mt. Pleasant, South Carolina
  - Memphis, Tennessee
  - Bellaire, Texas
  - Dallas, Texas
  - Denton, Texas
  - Houston, Texas
  - Burlington, Vermont
  - Charlottesville, Virginia
  - Richmond, Virginia
  - Morgantown, West Virginia
  - Middleton, Wisconsin
- Argentina (3):
  - Buenos Aires
  - La Plata
  - Mendoza
- Santiago, Chile
- Colombia (3):
  - Barranquilla
  - Bogotá
  - Bucamaranga
- Mexico (3):
  - Mexico City
  - Monterrey
  - Tobasco
- Peru (2):
  - Chiclayo
  - Lima

REFERENCES:
- [Derived] Soares CN, Thase ME, Clayton A, Guico-Pabia CJ, Focht K, Jiang Q, Kornstein SG, Ninan PT, Kane CP. Open-label treatment with desvenlafaxine in postmenopausal women with major depressive disorder not responding to acute treatment with desvenlafaxine or escitalopram. CNS Drugs. 2011 Mar;25(3):227-38. doi: 10.2165/11586460-000000000-00000. PMID 21323394

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in Argentina, Chile, Colombia, Mexico and the United States from December 2006 to January 2008.
Pre-assignment Details: Subjects were screened up to 4 weeks.
Groups:
- Desvenlafaxine Succinate Sustained-release (DVS SR): Acute Double Blind (DB) Phase Days 1 to 7: DVS SR 50 mg/day Days 8 to 14: 100 mg/day Days 15 to 56: At the discretion of the investigator, patients assigned 100 mg/day or 200 mg/day 6-Month Continuation Phases Double Blind Continuation Phase for Responders (HAM-D17 improved ≥50% from baseline) Days 57-238: continue taking DVS SR 100 mg/day or 200 mg/day Open-Label (OL) Extension Phase for Non-Responders (HAM-D17 improved <50% from baseline) Days 57-63: DVS SR 100 mg/day Days 64-238: At the discretion of the investigator, patients assigned DVS SR 100 mg/day or 200mg/day Taper Phase Day 239 or at discontinuation: If patient taking DVS SR 200 mg/day, then decreased to 100 mg for 7 days, and then decreased to 50 mg/day for 7 days. Patients taking DVS SR 100 mg/day decreased to 50 mg/day for 7 days.
- Escitalopram: Acute DB Phase Days 1-14:escitalopram 10mg/day; Days 15-56:discretion of the investigator patients assigned escitalopram 10mg/day or 20mg/day 6-Month Continuation Phases DB Continuation Phase for Responders (HAM-D17 improved > 50% from baseline) Days 57-238:continue taking escitalopram 10mg/day or 20mg/day OL Extension Phase for Non-Responders (HAM-D17 improved <50% from baseline) Days 57-63:DVS SR 100mg/day; Days 64-238:At the discretion of the investigator, patients assigned DVS SR 100mg/day or 200mg/day Taper Phase Day 239 or at discontinuation:If patient taking DVS SR 200mg/day, decreased to 100mg/day for 7 days, and then decreased to 50mg/day for 7 days. Patients taking DVS SR 100mg/day decreased to 50mg/day for 7 days. If patients taking escitalopram 20mg/day, decreased to 10mg/day for 7 days and then decreased to matching escitalopram placebo/day for 7 days. Patients taking escitalopram 10mg/day decreased to matching escitalopram placebo/day for 7 days.
Period: Acute Phase
Arm/Group | Desvenlafaxine Succinate Sustained-release (DVS SR) | Escitalopram
Started | 296 | 299
Completed | 245 | 256
Not Completed | 51 | 43
Not completed — Adverse Event | 18 | 13
Not completed — Failed to Return | 5 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 7 | 4
Not completed — Protocol deviation | 4 | 10
Not completed — Protocol Violation | 3 | 2
Not completed — Withdrawal by Subject | 11 | 9
Not completed — Lack of Efficacy | 3 | 3
Period: DB Continuation Phase for Responders
Arm/Group | Desvenlafaxine Succinate Sustained-release (DVS SR) | Escitalopram
Started | 172 | 188
Completed | 139 | 151
Not Completed | 33 | 37
Not completed — Adverse Event | 11 | 11
Not completed — Death | 1 | 0
Not completed — Failed to Return | 0 | 2
Not completed — Physician Decision | 2 | 3
Not completed — Lost to Follow-up | 1 | 7
Not completed — non-compliance | 7 | 5
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 8 | 6
Not completed — Lack of Efficacy | 1 | 1
Period: OL Extension Phase for Non-Responders
Arm/Group | Desvenlafaxine Succinate Sustained-release (DVS SR) | Escitalopram
Started | 69 | 60
Completed | 47 | 36
Not Completed | 22 | 24
Not completed — Adverse Event | 6 | 6
Not completed — Failed to Return | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 2 | 3
Not completed — non-compliance | 3 | 2
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Lack of Efficacy | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Desvenlafaxine Succinate Sustained-release (DVS SR) | Escitalopram | Total
Number analyzed (Participants) | 296 | 299 | 595
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.78 (6.13) | 56.15 (6.25) | 55.97 (6.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 296 | 299 | 595
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 211 | 219 | 430
  Mexico | 10 | 9 | 19
  Argentina | 43 | 42 | 85
  Chile | 11 | 9 | 20
  Colombia | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Psychiatric Rating Scale for Depression (HAM-D17) Score From Baseline to Week 8
Description: HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Items are scored on either a 3 point (0 to 2) or a 5 point scale (0 to 4) with 0=none/absent and 4=most severe,for a maximum total score of 50. Change= 8 week adjusted mean HAM-D17 minus baseline adjusted mean HAM-D17.
Time Frame: Baseline and 8 weeks
Population: Acute Double-blind phase; all randomized patients with a baseline HAM-D17 score ≥ 18, who took at least 1 dose of study drug and had at least 1 post-baseline HAM-D17 evaluation.
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Desvenlafaxine Succinate Sustained-release (DVS SR) | Escitalopram
Number analyzed (Participants) | 185 | 203
units on scale | -13.63 (0.42) | -14.30 (0.40)
Statistical Analysis 1: Comparison: Desvenlafaxine Succinate Sustained-release (DVS SR) vs Escitalopram; DVS SR compared with ESC; Test type: Superiority or Other; p = 0.243, Mixed Models Analysis; Mixed Models Repeated Measures (MMRM) with baseline score as a covariant and factors for center, week and treatment; Mean Difference (Final Values) = 0.67, 95% CI [-0.46 to 1.81] — DVS SR adjusted mean change minus ESC adjusted mean change

2. Secondary Outcome: Percentage of Patients Achieving Response to Treatment at Final On-therapy Evaluation (Acute Phase)
Description: A response is defined as ≥ 50% decrease from baseline on Hamilton Psychiatric Rating Scale for Depression (HAM-D17) score. HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Individual items are scored on a 0 to 2 or 4 scale (0=none/absent and 4=most severe) for a maximum total score of 50.
Time Frame: 8 weeks
Population: Acute double-blind phase; all randomized patients with a baseline HAM-D17 score ≥18, who took at least 1 dose of study drug and had at least 1 post-baseline HAM-D17 evaluation.
Measure: Number; unit: percentage of patients
Arm/Group | Desvenlafaxine Succinate Sustained-release (DVS SR) | Escitalopram
Number analyzed (Participants) | 224 | 237
percentage of patients | 64.3 | 73.4
Statistical Analysis 1: Comparison: Desvenlafaxine Succinate Sustained-release (DVS SR) vs Escitalopram; DVS SR compared with ESC; Test type: Superiority or Other; p = 0.077, Chi-squared; Logistic regression model with treatment and site as factors and baseline score as a covariant; Odds Ratio (OR) = 0.608, 95% CI [0.40 to 0.92] — Estimated odds ratio of DVS SR to ESC. Odd ratio adjusted for baseline, treatment and site

3. Secondary Outcome: Percentage of Patients Achieving Remission at Final On-therapy Evaluation (Acute Phase)
Description: Remission is defined as a Hamilton Psychiatric Rating Scale for Depression (HAM-D17) score of ≤ 7. HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Individual items are scored on a 0 to 2 or 4 scale (0=none/absent and 4=most severe) for a maximum total score of 50.
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of patients
Arm/Group | Desvenlafaxine Succinate Sustained-release (DVS SR) | Escitalopram
Number analyzed (Participants) | 224 | 237
Percentage of patients | 37.9 | 48.1
Statistical Analysis 1: Comparison: Desvenlafaxine Succinate Sustained-release (DVS SR) vs Escitalopram; DVS SR compared with ESC; Test type: Superiority or Other; p = 0.0054, Chi-squared; Logistic regression model with treatment and site as factors and baseline score as a covariant; Odds Ratio (OR) = 0.571, 95% CI [0.39 to 0.85] — Estimated odds ratio of DVS SR to ESC. Odds ratio adjusted for baseline, treatment and site

4. Secondary Outcome: Clinical Global Impression Improvement (CGI-I) Score at 8 Weeks
Description: CGI-I is a global rating scale that measures disease improvement. Using a 7-point scale, the clinician rates how much the patient's illness has improved or worsened relative to the baseline status (1= very much improved; 7= very much worse).
Time Frame: 8 weeks
Population: Acute double-blind phase; all randomized patients with a baseline HAM-D17 score ≥18, took at least1 dose of study drug and had at least1 post-baseline HAM-D17 evaluation.
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Desvenlafaxine Succinate Sustained-release (DVS SR) | Escitalopram
Number analyzed (Participants) | 185 | 203
units on scale | 1.93 (0.08) | 1.81 (0.07)
Statistical Analysis 1: Comparison: Desvenlafaxine Succinate Sustained-release (DVS SR) vs Escitalopram; DVS SR compared with ESC; Test type: Superiority or Other; p = 0.260, Mixed Models Analysis; Mixed Models Repeated Measures (MMRM) with baseline score as a covariant and factors for center, week and treatment; Mean Difference (Final Values) = 0.12, 95% CI [-0.09 to 0.33] — DVS SR minus ESC adjusted mean

5. Secondary Outcome: Change in Clinical Global Impression Severity (CGI-S) Score From Baseline to Week
Description: CGI-S is a global rating scale that measures the severity of a patient's disease. Using a 7-point scale, the clinician rates the severity of the patient's mental illness at the time of the assessment, relative to the clinician's experience with patients who have the same diagnosis (1= normal; 7= extremely ill).
Time Frame: Baseline and 8 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Desvenlafaxine Succinate Sustained-release (DVS SR) | Escitalopram
Number analyzed (Participants) | 185 | 203
units on scale | -2.09 (0.09) | -2.22 (0.08)
Statistical Analysis 1: Comparison: Desvenlafaxine Succinate Sustained-release (DVS SR) vs Escitalopram; Test type: Superiority or Other; p = 0.239, Mixed Models Analysis; Mixed Models Repeated Measures (MMRM) with baseline score as a covariant and factors for center, week and treatment; Mean Difference (Final Values) = 0.14, 95% CI [-0.09 to 0.37] — DVS SR minus ESC adjusted mean

6. Secondary Outcome: Change in Hamilton Psychiatric Rating Scale for Anxiety From Baseline to Week 8 (HAM-A) Score
Description: The HAM-A is a standardized, clinician-administered rating scale that assesses 14 items characteristically associated with major anxiety disorders. Items are scaled 0 - 4 (0=none and 4=very severe), with a maximum total score of 56. Change= 8 week adjusted mean HAM-A total score minus baseline adjusted mean total score.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Desvenlafaxine Succinate Sustained-release (DVS SR) | Escitalopram
Number analyzed (Participants) | 185 | 203
units on scale | -11.37 (0.42) | -11.73 (0.40)
Statistical Analysis 1: Comparison: Desvenlafaxine Succinate Sustained-release (DVS SR) vs Escitalopram; DVS SR compared to ESC; Test type: Superiority or Other; p = 0.516, Mixed Models Analysis; Mixed model Repeated Measures (MMRM) analysis adjusted mean score for baseline score, time and center; Mean Difference (Net) = 0.37, 95% CI [-0.75 to 1.49] — DVS SR adjusted mean change minus ESC adjusted mean change

7. Secondary Outcome: Change in Dimension Health State EuroQol (EQ-5D) Score From Baseline to Week 8
Description: EQ-5D is a standardized, subject-administered measure of health outcome. It provides a descriptive profile for 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), using 3 levels (no, moderate, or extreme problems) and a single index value characterizing current health status using a 100-point visual analog scale (0=worst, 100=best). EQ-5D summary index is obtained with a formula that weights each level of the dimensions. The index-based score is interpreted along a continuum of 0 (death) to 1 (perfect health). Change=8 week score minus baseline score.
Time Frame: Baseline and week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Desvenlafaxine Succinate Sustained-release (DVS SR) | Escitalopram
Number analyzed (Participants) | 179 | 189
units on scale | 0.25 (0.02) | 0.24 (0.02)
Statistical Analysis 1: Comparison: Desvenlafaxine Succinate Sustained-release (DVS SR) vs Escitalopram; DVS SR compared to ESC; Test type: Superiority or Other; p = 0.635, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM) with treatment, time and site as factors and baseline as covariant; Mean Difference (Net) = 0.01, 95% CI [-0.03 to 0.06] — DVS SR adjusted mean change minus ESC adjusted mean change

8. Secondary Outcome: Percentage of Responders Maintaining Response to Treatment at Final On-therapy Evaluation (Double Blind Continuation Phase)
Description: Patients achieving a response to treatment at the end of the 8-week acute double blind (DB) phase continued the same treatment in a 6-month DB continuation phase and were evaluated to see if the response was maintained. A response is defined as ≥ 50% decrease from baseline on Hamilton Psychiatric Rating Scale for Depression (HAM-D17) score. HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Individual items are scored on a 0 to 2 or 4 scale (0=none/absent and 4=most severe) for a maximum total score of 50.
Time Frame: 6 months
Population: All randomized patients with a baseline HAM-D17 score ≥18, who took at least 1 dose of study drug, had at least 1 post-baseline HAM-D17 evaluation, achieved a response to treatment (≥50% reduction of HAM-D17 total score from baseline) at the end of the acute phase (week 8) and continued treatment in the double blind continuation phase.
Measure: Number; unit: percentage of responders
Groups:
- DVS SR Responders / DVS SR DB: Patients who received DVS SR during the acute double blind phase (weeks 1-8), achieved a response to treatment (defined as HAM-D17 improved ≥50% from baseline) at the end of the acute phase and continued on DVS SR during the 6-month Double Blind Continuation phase.
- ESC Responders / ESC DB: Patients who received ESC during the acute double blind phase (weeks 1-8), achieved a response to treatment (defined as HAM-D17 improved ≥50% from baseline) at the end of the acute phase and continued on ESC during the 6-month Double Blind Continuation phase.
Arm/Group | DVS SR Responders / DVS SR DB | ESC Responders / ESC DB
Number analyzed (Participants) | 137 | 160
percentage of responders | 81.8 | 80.0
Statistical Analysis 1: Comparison: DVS SR Responders / DVS SR DB vs ESC Responders / ESC DB; DVS SR compared with ESC; Test type: Superiority or Other; p = 0.702, Chi-squared; Odds Ratio (OR) = 1.12, 95% CI [0.63 to 2.00] — Estimated odds ratio of DVS SR to ESC. Odd ratio adjusted for baseline, treatment and site

9. Secondary Outcome: Percentage of Responders Achieving Remission at Final On-therapy Evaluation (Double Blind Continuation Phase)
Description: Patients achieving a response to treatment at the end of the 8-week acute double blind (DB) phase continued the same treatment in a 6-month DB continuation phase and were evaluated to see if remission was achieved. Remission is defined as a Hamilton Psychiatric Rating Scale for Depression (HAM-D17) score of ≤ 7. HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Individual items are scored on a 0 to 2 or 4 scale (0=none/absent and 4=most severe) for a maximum total score of 50.
Time Frame: 6 months
Population: as for outcome 8
Measure: Number; unit: percentage of responders
Arm/Group | DVS SR Responders / DVS SR DB | ESC Responders / ESC DB
Number analyzed (Participants) | 137 | 160
percentage of responders | 67.9 | 61.3
Statistical Analysis 1: Comparison: DVS SR Responders / DVS SR DB vs ESC Responders / ESC DB; DVS SR compared with ESC; Test type: Superiority or Other; p = 0.234, Chi-squared; Odds Ratio (OR) = 1.34, 95% CI [0.83 to 2.16] — Estimated odds ratio of DVS SR to ESC. Odd ratio adjusted for baseline, treatment and site

10. Secondary Outcome: Percentage of Responders Improving Response to Remission During 6-month Double Blind Continuation Phase
Description: Patients achieving a response to treatment (Responders) at the end of the 8-week acute double blind (DB) phase continued into a 6-month DB phase. Responders without remission at 8 weeks were assessed for remission status during the 6-month continuation. Remission defined as a Hamilton Psychiatric Rating Scale for Depression (HAM-D17) score ≤ 7. HAM-D17 is a standardized, clinician-administered rating scale assessing 17 items characteristically associated with major depression. Individual items scored on a 0 to 2 or 4 scale (0=none/absent and 4=most severe) for a maximum total score of 50.
Time Frame: 6 months
Population: All randomized patients with baseline HAM-D17 score ≥18, who took ≥1 dose study drug, had ≥1 post-baseline HAM-D17 evaluation, achieved a response to treatment (≥50% reduction of HAM-D17 total score from baseline) but not remission (HAM-D17 score ≤ 7) at the end of the acute phase and continued treatment in the 6-month DB continuation phase.
Measure: Number; unit: percentage of responders
Arm/Group | DVS SR Responders / DVS SR DB | ESC Responders / ESC DB
Number analyzed (Participants) | 54 | 55
percentage of responders | 88.9 | 81.8

11. Secondary Outcome: Percentage of Non-Responders Achieving Response at Final Evaluation of 6-month Open-Label (OL)Extension Phase
Description: Patients who didn't achieve a response to treatment at the end of the 8-week acute double blind phase entered into an OL treatment phase with DVS SR for 6 months and were evaluated to see if a response was achieved. A response is defined as ≥ 50% decrease from baseline on Hamilton Psychiatric Rating Scale for Depression (HAM-D17) score. HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Individual items are scored on a 0 to 2 or 4 scale (0=none/absent and 4=most severe) for a maximum total score of 50.
Time Frame: 6 months
Population: All randomized patients who took at least 1 dose of study drug, who did not achieve a response to treatment (≥50% reduction of HAM-D17 total score from baseline) at the end of the acute phase (week 8), entered into the open label extension phase and had baseline and at least 1 post-baseline HAM-D17 evaluation in the acute and open label phase.
Measure: Number; unit: Percentage of Non-Responders
Groups:
- DVS SR Non-Responders / DVS SR OL: Patients who received DVS SR during the acute double blind phase (weeks 1-8), did not achieve a response to treatment (response defined as HAM-D17 improved ≥50% from baseline) at the end of the acute phase; entered into open label (OL) treatment with DVS SR during 6-month Open Label Extension phase.
- ESC Non-Responders / DVS SR OL: Patients who received ESC during the acute double blind phase (weeks 1-8), did not achieve a response to treatment (response defined as HAM-D17 improved ≥50% from baseline) at the end of the acute phase; entered into open label (OL) treatment with DVS SR during 6-month Open Label Extension phase.
Arm/Group | DVS SR Non-Responders / DVS SR OL | ESC Non-Responders / DVS SR OL
Number analyzed (Participants) | 185 | 203
Percentage of Non-Responders | 39.1 | 50.8

12. Secondary Outcome: Percentage of Non-Responders Achieving Remission at Final Evaluation of 6-month Open-Label Extension Phase
Description: Patients who did not achieve a response to treatment at the end of the 8-week acute double blind phase entered into an open label (OL) treatment phase with DVS SR for 6 months and were evaluated to see if remission was achieved. Remission is defined as a Hamilton Psychiatric Rating Scale for Depression (HAM-D17) score of ≤ 7. HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Individual items are scored on a 0 to 2 or 4 scale (0=none/absent and 4=most severe) for a maximum total score of 50.
Time Frame: 6 months
Population: as for outcome 11
Measure: Number; unit: Percentage of Non-Responders
Arm/Group | DVS SR Non-Responders / DVS SR OL | ESC Non-Responders / DVS SR OL
Number analyzed (Participants) | 64 | 59
Percentage of Non-Responders | 40.6 | 47.5

13. Secondary Outcome: Discontinuation-Emergent Signs and Symptoms (DESS) Total Score
Description: DESS is a clinician-administered 43-item assessment that evaluates discontinuation-emergent symptoms resulting from the withdrawal from test article. The DESS total score is the sum of the number of new symptoms and old (but worse) symptoms that appeared during tapering of the test article. A higher score indicates more symptoms. The DESS score was assessed by status of taper.
Time Frame: 6 months
Population: Safety population: Randomized patients who took ≥1 dose study drug. Excluded patients lost to follow-up and discontinued with < 4 wks therapy. Patients analyzed varied by time (DVS SR, ESC): End of Therapy (n=264, 267); Taper week 1 (n=217, 227); Taper week 2 (n=222, 223); Post-taper (n=219, 223).
Measure: Mean (Standard Deviation); unit: units on scale
Groups:
- Desvenlafaxine Succinate Sustained-Release (DVS SR): Taper Phase Day 239 or at discontinuation: If patient taking DVS SR 200 mg/day, then decreased to 100 mg/day for 7 days, and then decreased to 50 mg/day for 7 days. Patients taking DVS SR 100 mg/day decreased to 50 mg/day for 7 days.
- Escitalopram (ESC): Taper Phase Day 239 or at discontinuation: If patients taking escitalopram 20 mg/day, then decrease to 10 mg/day for 7 days and then decreased to matching escitalopram placebo/day for 7 days. Patients taking escitalopram 10 mg/day decreased to matching escitalopram placebo/day for 7 days.
Arm/Group | Desvenlafaxine Succinate Sustained-Release (DVS SR) | Escitalopram (ESC)
Number analyzed (Participants) | 264 | 267
units on scale
  End of Therapy | 1.49 (3.09) | 1.52 (3.65)
  Taper week 1 | 1.18 (2.12) | 1.68 (3.28)
  Taper week 2 | 2.29 (3.46) | 3.16 (4.58)
  Post-taper | 1.61 (3.55) | 1.48 (2.86)
Statistical Analysis 1: Comparison: Desvenlafaxine Succinate Sustained-Release (DVS SR) vs Escitalopram (ESC); DVS SR vs. ESC: end of therapy; Test type: Superiority or Other; p = 0.927, t-test, 2 sided
Statistical Analysis 2: Comparison: Desvenlafaxine Succinate Sustained-Release (DVS SR) vs Escitalopram (ESC); DVS SR vs. ESC: after 1 week of taper; Test type: Superiority or Other; p = 0.055, t-test, 2 sided
Statistical Analysis 3: Comparison: Desvenlafaxine Succinate Sustained-Release (DVS SR) vs Escitalopram (ESC); DVS SR vs. ESC: after 2 weeks of taper; Test type: Superiority or Other; p = 0.025, t-test, 2 sided
Statistical Analysis 4: Comparison: Desvenlafaxine Succinate Sustained-Release (DVS SR) vs Escitalopram (ESC); DVS SR vs. ESC: after > 2 weeks of taper; Test type: Superiority or Other; p = 0.653, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Desvenlafaxine Succinate Sustained-release (DVS SR) | Escitalopram
Serious Adverse Events (participants affected / at risk) | 5 | 4
Other Adverse Events (participants affected / at risk) | 267 | 262
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Desvenlafaxine Succinate Sustained-release (DVS SR) | Escitalopram
Accidental injury (General disorders) | 0/296 | 1/299
Non-specific drug reaction (General disorders) | 1/296 | 0/299
Overdose (General disorders) | 0/296 | 1/299
Suicide attempt (General disorders) | 2/296 | 0/299
Postural hypotension (Cardiac disorders) | 1/296 | 0/299
Hepatitis (Hepatobiliary disorders) | 1/296 | 0/299
Hepatomegaly (Hepatobiliary disorders) | 1/296 | 0/299
Anxiety (Nervous system disorders) | 1/296 | 0/299
Depression (Nervous system disorders) | 1/296 | 1/299
Hypesthesia (Nervous system disorders) | 0/296 | 1/299
Paresis (Nervous system disorders) | 0/296 | 1/299
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Desvenlafaxine Succinate Sustained-release (DVS SR) | Escitalopram
Abdominal pain (General disorders) | 29/296 | 21/299
Asthenia (General disorders) | 27/296 | 23/299
Back pain (General disorders) | 16/296 | 13/299
Headache (General disorders) | 76/296 | 85/299
Infection (General disorders) | 17/296 | 21/299
Hypertension (Cardiac disorders) | 16/296 | 15/299
Vasodilatation (Vascular disorders) | 12/296 | 16/299
Anorexia (Gastrointestinal disorders) | 20/296 | 15/299
Constipation (Gastrointestinal disorders) | 52/296 | 28/299
Diarrhea (Gastrointestinal disorders) | 26/296 | 49/299
Dry mouth (Gastrointestinal disorders) | 83/296 | 60/299
Dyspepsia (Gastrointestinal disorders) | 21/296 | 27/299
Nausea (Gastrointestinal disorders) | 74/296 | 61/299
Metabolic and nutritional (Metabolism and nutrition disorders) | 20/296 | 13/299
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 26/296 | 32/299
Dizziness (Nervous system disorders) | 33/296 | 28/299
Insomina (Nervous system disorders) | 33/296 | 39/299
Nervousness (Nervous system disorders) | 21/296 | 10/299
Sommolence (Nervous system disorders) | 42/296 | 48/299
Respiratory (Respiratory, thoracic and mediastinal disorders) | 29/296 | 28/299
Sweating (Skin and subcutaneous tissue disorders) | 43/296 | 33/299
Abnormal vision (Eye disorders) | 14/296 | 17/299
Urogenitial (Renal and urinary disorders) | 24/296 | 25/299

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.